CLINICAL TRIAL: NCT01055145
Title: Comparison of the Effect Between Levofloxacin and Moxifloxacin on the Culture Conversion After 3 Months Treatment Among MDR-TB Patients; Prospective Multicenter Randomized Open Label Phase III Trial
Brief Title: Comparison of the Effect Between Levofloxacin and Moxifloxacin Among MDR-TB Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Jae-Joon Yim / Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-0911-068-301
Record Dates: First submitted 2010-01-21; First posted 2010-01-25 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: TB
Keywords: Multidrug-resistant TB, sensitive to levofloxacin and moxifloxacin
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant | interventions — Levofloxacin; Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- levofloxacin (Active Comparator): Levofloxacin 750mg po per day for 3 months
  Interventions: Drug: levofloxacin, moxifloxacin
- moxifloxacin (Active Comparator): Moxifloxacin 400mg po per day for 3 months
  Interventions: Drug: levofloxacin, moxifloxacin

INTERVENTIONS:
Drug: levofloxacin, moxifloxacin — Levofloxacin 750mg po per day for 3 months vs. Moxifloxacin 400mg po per day for 3 months

SUMMARY:
Fluoroquinolone is a one of the most important drugs for treatment of multidrug-resistant TB (MDR-TB). Among them, levofloxacin and moxifloxacin has been used most widely. However, there is no study to directly compare the efficacy of levofloxacin and moxifloxacin among MDR-TB patients. The investigators will compare the efficacy of levofloxacin and moxifloxacin through a prospective multicenter randomized open label phase III trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multidrug-resistant TB, but sensitive to levofloxacin and moxifloxacin

Exclusion Criteria:

* Achieved negative conversion of M. TB culture before the enrollment
* Positive anti-HIV antibody
* Pregnant women or sexually active women without using proper birth control method
* Serum creatine grater than 2mg/dL, or urine protein greater than 2+
* Serum total bilirubin greater than 2 mg/dL or AST and ALT greater than 1.5 times of normal upper limit
* History or current arrhythmia
* Hypersensitivity to levofloxacin, moxifloxacin,or rifabutin
* Should use drug containing metal-ion, warfarin, phenytoin, theophylline, probenecid regularly

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2010-03; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Negative conversion of M. tuberculosis | 3 months after initiation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Joon Yim, MD, Principal Investigator — Seoul National University Hospital
Locations (29):
- South Korea (29):
  - Korea University Ansan Hospital, Ansan, Gyeonggi-do
  - Catholic University of Korea Bucheon St. Mary's Hospital, Bucheon-si, Gyeonggi-do
  - Bundang CHA Hospital, Bundang, Gyeonggi-do
  - Seoul National University Bundang Hospital, Bundang, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Pyeongchon, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Seoul National University Hospital, Seoul, Seoul
  - Kangwon National University Hospital, Chuncheon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Hospital, Incheon
  - Gyeongsang National University Hospital, Jinju
  - Masan Samsung Medical Center, Masan
  - Inje University Pusan Paik Hospital, Pusan
  - Pusan National University Hospital, Pusan
  - Asan Medical Center, Seoul
  - Chung-Ang University Yong-san Hospital, Seoul
  - East-West Neo Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Inje University Sanggye Paik Hospital, Seoul
  - Kangbuk Samsung Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Korean Institute of Tuberculosis, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Medical Center, Seoul
  - Seoul National University Boramae Medical Center, Seoul
  - Severance Hospital, Seoul

REFERENCES:
- [Derived] Kang YA, Shim TS, Koh WJ, Lee SH, Lee CH, Choi JC, Lee JH, Jang SH, Yoo KH, Jung KH, Kim KU, Choi SB, Ryu YJ, Kim KC, Um S, Kwon YS, Kim YH, Choi WI, Jeon K, Hwang YI, Kim SJ, Lee HK, Heo E, Yim JJ. Choice between Levofloxacin and Moxifloxacin and Multidrug-Resistant Tuberculosis Treatment Outcomes. Ann Am Thorac Soc. 2016 Mar;13(3):364-70. doi: 10.1513/AnnalsATS.201510-690BC. PMID 26871879
- [Derived] Koh WJ, Lee SH, Kang YA, Lee CH, Choi JC, Lee JH, Jang SH, Yoo KH, Jung KH, Kim KU, Choi SB, Ryu YJ, Chan Kim K, Um S, Kwon YS, Kim YH, Choi WI, Jeon K, Hwang YI, Kim SJ, Lee YS, Heo EY, Lee J, Ki YW, Shim TS, Yim JJ. Comparison of levofloxacin versus moxifloxacin for multidrug-resistant tuberculosis. Am J Respir Crit Care Med. 2013 Oct 1;188(7):858-64. doi: 10.1164/rccm.201303-0604OC. PMID 23927582